CLINICAL TRIAL: NCT06181214
Title: The Effects of a Novel Nutritional Product on Nutrient Status and Digestive Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Athletic Greens International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: AG-01-0623
Record Dates: First submitted 2023-12-05; First posted 2023-12-26 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Gastrointestinal Microbiome; Nutrition, Healthy; Healthy Aging

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo Controlled Design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Maltodextrin + Flavoring
  Interventions: Dietary Supplement: Placebo
- AG1 - Nutritional Supplement (Experimental): A foundational nutritional supplement consisting of vitamins, minerals, probiotics, prebiotics, and whole food ingredients
  Interventions: Dietary Supplement: AG1 - Nutritional Supplement

INTERVENTIONS:
Dietary Supplement: AG1 - Nutritional Supplement — A foundational nutritional supplement consisting of vitamins, minerals, probiotics, prebiotics, and whole food ingredients
  Arms: AG1 - Nutritional Supplement
Dietary Supplement: Placebo — Maltodextrin placebo
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled study of N=30 apparently healthy men and women. This is an exploratory study to assess the effect of a novel dietary supplement on blood markers of nutrient status and the gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Provide voluntary signed and dated informed consent.
* Be in good health as determined by medical history and routine blood chemistries.
* Age between 18 and 50 yr (inclusive).
* Body Mass Index of 18.5-29.9 (inclusive).
* Body weight of at least 120 pounds.
* Normotensive (seated, resting systolic blood pressure <140 mm Hg and diastolic blood pressure < 90 mm Hg. If the first measurement is slightly elevated above these limits, the subject will be given a brief (5 minute) rest period, and two more measurements will be taken. The average of all three measurements will be used to determine eligibility.
* Normal seated, resting heart rate (<90 per minute).
* Willing to duplicate their previous 24-hour diet, refrain from caffeine and exercise for 24 hours prior to each visit, and fast for 10 hours prior to each visit.
* Subject agrees to maintain existing dietary and physical activity patterns throughout the study period.
* Subject is willing and able to comply with the study protocol.

Exclusion Criteria:

* History of unstable or new-onset cardiovascular/cardiorespiratory, liver, or renal conditions.
* History of diabetes or endocrine disorder.
* History of use of medications or dietary supplements known to confound the study or its endpoints.
* Alcohol consumption (more than 2 standard alcoholic drinks per day or more than 10 drinks per week) or drug abuse or dependence within the past 6 months.
* Current smokers or smoking within the past month.
* History of hyperparathyroidism or an untreated thyroid condition.
* History of malignancy in the previous 5 years except for non-melanoma skin cancer (basal cell cancer or squamous cell cancer of the skin).
* Prior gastrointestinal bypass surgery (Lapband), etc.
* Other known gastrointestinal or metabolic conditions that might impact nutrient absorption or metabolism, e.g., short bowel syndrome, Irritable bowel syndrome (IBS), diarrheal illnesses, history of colon resection, gastro paresis, Inborn-Errors-of-Metabolism (such as PKU).
* Chronic inflammatory condition (e.g., rheumatoid arthritis, Crohn's, ulcerative colitis, Lupus, HIV/AIDS, etc.).
* Previous medical diagnosis of asthma, gout, or fibromyalgia.
* Pregnant women, women trying to become pregnant, women less than 120 days postpartum or nursing women. Women who participate in this study must agree to the use of contraception for the duration of the study and any woman that is sexually active will have to take a negative pregnancy test prior to enrolling. Women of childbearing age (any woman prior to menopause) regardless of their use of contraception will be provided a urine pregnancy test kit at their screening visit and take the test in private using the female lavatory after signing an informed consent.
* Known sensitivity to any ingredient in the test formulations as listed in the product label.
* Currently participating in another research study with an investigational product or have been in another research study in the past 30 days.
* Any other conditions that, in the opinion of the medical staff, could confound the primary endpoints or place the subject at increased risk of harm if they were to participate.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Gut Microbiome | 28 days
  Examine changes in the gut microbiome structure and function measured by shallow shotgun metagenomics. Examine enrichment of taxa and metabolic pathways in the gut microbiome as a result of dietary supplementation.

SECONDARY OUTCOMES:
Complete Metabolic Blood Panel | 28 Days
  Serum concentrations of sodium, potassium, carbon dioxide, chloride, albumin, total protein, glucose, and calcium., ALT, AST, bilirubin, BUN, creatinine
Complete Blood Count | 28 Days
  Circulating concentrations of white blood cells, red blood cells, hemoglobin, and hematocrit
Exploratory nutrient status markers | 28 days
  Circulating concentrations of nutrient status (e.gg, zinc, vitamin c, folate, & magnesium)
Exploratory Digestive Measures | 28 days
  A Digestive Quality of Life Questionnaire (DQLQ) will be utilized to assess the effect of the interventions on participant's digestive health. Scores range from 0 to 9 with a higher score indicating worse digestion associated with quality of life
Exploratory Stool Consistency | 28 days
  Bristol Stool Scale (score 1-7) questionnaire that allows participants to identify how loose or hard their stool consistency is
Exploratory Stool Frequency | 28 days
  100mm Visual Analog Scale (VAS) to assess subjective ratings of stool consistency and frequency of bowl movements

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Applied Health Sciences, Canfield, Ohio, United States

REFERENCES:
- [Derived] La Monica MB, Raub B, Hartshorn S, Gustat AL, Grdic J, Kirby TO, Townsend JR, Sandrock J, Ziegenfuss TN. The effects of AG1(R) supplementation on the gut microbiome of healthy adults: a randomized, double-blind, placebo-controlled clinical trial. J Int Soc Sports Nutr. 2024 Dec;21(1):2409682. doi: 10.1080/15502783.2024.2409682. Epub 2024 Oct 1. PMID 39352252